CLINICAL TRIAL: NCT02599285
Title: Operative Treatment of AO Weber C Fibular Fractures With Additional Medium-sized Posterior Malleolar Fragment: Syndesmotic Reduction and Functional Outcome After Syndesmotic Positioning Screws or Posterior Fragment Fixation. POSTFIX-C Trial: a Prospective Comparative Observational Study.
Brief Title: Fixation of the Posterior Malleolus in Trimalleolar AO Weber C Fractures.
Acronym: POSTFIX-C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Center Haaglanden (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Jochem Hoogendoorn, Dr., Medical Center Haaglanden
Other Study IDs: NL50169.098.15
Record Dates: First submitted 2015-11-03; First posted 2015-11-06 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Trimalleolar Fracture; AO Weber C Fractures; Syndesmotic Stability; Open Reduction and Internal Fixation
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fixation: Patients with a trimalleolar AO Weber C fracture with open reduction and fixation of the posterior malleolar fragment.
  Interventions: Device: Fixation
- No Fixation: Patients with a trimalleolar AO Weber C fracture without open reduction and fixation of the posterior malleolar fragment.
  Interventions: Device: NO Fixation

INTERVENTIONS:
Device: Fixation — Fixation of the posterior malleolus with lag-screws or plate-fixation. If syndesmosis is intra-operatively stable, no syndesmotic positioning screws will be placed.
  Groups: Fixation
Device: NO Fixation — Posterior malleolus will not be fixated. Syndesmotic positioning screws will be placed.
  Groups: No Fixation

SUMMARY:
In AO Weber type C fractures, there is a combination of a proximal fibular fracture, a medial fracture or ruptured deltoid ligament, and a syndesmotic injury. Anatomical repair and reduction of the syndesmosis is essential to prevent diastasis in the ankle-joint. Widening and chronical instability of the syndesmosis is related to worse functional outcome and development of posttraumatic osteoarthritis in the ankle. There is limited biomechanical and clinical evidence that syndesmotic stability in AO Weber type C fractures with an additional posterior malleolar fracture can also be reached by fixation of the posterior malleolar fragment. Maybe, this is even superior to the usual treatment with syndesmotic positioning screws. Some authors concluded that stability of the syndesmosis in these fractures can be much more achieved by fixation of the posterior malleolar fragment than by placement of syndesmotic positioning screws alone. Another additional benefit of open reduction and fixation of the posterior malleolar fragment is that this will lead to an anatomical reconstruction of the syndesmosis. Although there is no current evidence, it is likely that a malreduction of the fibula in the tibial incisura will lead to a worse functional outcome on the long-term. No clear consensus in the literature is found as to which fragment size of the posterior malleolus should be internally fixed. The general opinion is that displaced fragments that involve more than 25% of the distal articular tibia should be fixed. Traditionally, reduction of these larger fragments is indirectly, followed by percutaneous screw fixation in anterior-posterior direction. Disadvantages are that it is hard to achieve an anatomical reduction, and that percutaneous fixation of smaller fragments is very difficult. Recently, a direct exposure of the posterior tibia via a posterolateral approach in prone position, followed by open reduction and fixation with screws in posterior-anterior direction or antiglide plate is advocated by several authors. This approach allows perfect visualization of the fracture, articular anatomical reduction, and strong fixation. Another advantage is that even small posterior fragments can be addressed. Several case series are published, which describe minimal major wound complications, good functional outcomes, and minimal need for reoperation.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years
2. First ankle fracture of the affected side
3. Isolated, fibular fracture proximal to the syndesmosis with a posterior malleolar fragment between 5 and 25% of the involved articular surface(AO type 44-C1, 44-C2, 44-C3).

Exclusion Criteria:

1. Multiple injuries
2. Ankle fracture of the same ankle in the history
3. Patients with pre-existent mobility problems
4. Pre-existent disability like wheelchair or walking aid dependency.
5. Patients living in another region of whom follow-up will take place in another hospital
6. Insufficient understanding of the Dutch language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with a trimalleolar AO-Weber C fracture with additional posterior fragment (5-25% of the involved articular surface, AO type 44-C1, 44-C2, 44-C3) in the participating hospitals between the age of 18 and 70 could be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2015-11; Primary Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of syndesmotic reduction 1cm above the tibial plafond, measured on post-operative CT-scan in millimeters compared to the contralateral (healthy) side. | 1 year
Functional outcome measured by AAOS score (special questionnaire for hindfoot and ankle in 27 questions.) | 1 Year

SECONDARY OUTCOMES:
Posttraumatic osteoarthritis defined by the Kellgren-Lawrence score (1-4) | 5 Years

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Leiden University Medical Center, Leiden, South Holland
  - MCHaaglanden, The Hague, South Holland
  - Bronovo Ziekenhuis, The Hague, South Holland
  - Haga ziekenhuis, The Hague, South Holland